CLINICAL TRIAL: NCT07250789
Title: Cognitive Screening of Individuals Diagnosed With Type 2 Diabetes and the Impact of a Multidomain Intervention Targeting Cognitive Decline (The Brain Care Study)
Brief Title: Cognitive Screening and Multidomain Intervention Targeting Cognitive Decline in Type 2 Diabetes (The Brain Care Study)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Steno Diabetes Center Copenhagen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H-24006680
Record Dates: First submitted 2025-11-18; First posted 2025-11-26 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Diabetes; Diabetes Mellitus Type 2; Type 2 Diabetes; Type 2 Diabetes Mellitus (T2DM); Cognitive Impairment; Cognitive Decline
Keywords: diabetes; type 2 diabetes; type 2 diabetes mellitus; t2d; t2dm; cognitive impairment; cognitive decline
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2; Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental)
  Interventions: Other: Multidomain Intervention Targeting Cognitive Decline
- Usual Care (No Intervention)

INTERVENTIONS:
Other: Multidomain Intervention Targeting Cognitive Decline — The multidomain intervention will include the following: Optimization of pharmacological treatment/Pharmacological neuroprotection. Adjustment of HbA1c targets. Vascular risk factor management. Assessment of hearing impairment. Assessment of depression. Dialogue tools. Social interaction. Guidance on physical training. Cognitive training. Text message reminders.
  Arms: Intervention

SUMMARY:
The purpose of The Brain Care Study is to investigate the prevalence of cognitive impairment in older adults with type 2 diabetes (T2D) and to evaluate the effectiveness of a multidomain intervention designed to prevent cognitive decline.

DETAILED DESCRIPTION:
Type 2 diabetes (T2D) is a chronic condition associated with cognitive decline and an increased risk of Alzheimer's disease and vascular dementia. Cognitive impairment in individuals with T2D complicates disease management, often leading to poorer clinical outcomes. Although guidelines recommend cognitive screening for older adults with T2D, uncertainties remain regarding how to best identify high-risk individuals and adjust treatment strategies. While multidomain interventions have shown potential in delaying cognitive decline, further research is needed to develop feasible and effective strategies for at-risk populations.

The Brain Care Study consists of two parts: a prevalence study involving cognitive screening and a two-year randomized controlled trial (RCT) to assess a multidomain intervention targeting multiple risk factors, including pharmacological optimization, lifestyle changes, and social interaction.

The multidomain intervention focuses on optimizing medication, adjusting HbA1c targets, managing vascular risk factors, and addressing hearing impairment, depression, physical activity, and cognitive training. Additionally, the study will employ dialogue tools, text message reminders, and social interaction to enhance participants' health and adherence to the intervention.

The study hypothesizes that cognitive screening will be feasible and will not increase diabetes-related distress, while the intervention may reduce cognitive decline, improve health-related quality of life, decrease hospitalization rates, and minimize the need for home visits or relocation to nursing homes. Study endpoints include the prevalence of cognitive impairment, changes in cognitive function, hospitalization rates, and medication adherence, with the goal of providing evidence-based recommendations for future diabetes care guidelines.

Overall, the Brain Care Study aims to quantify the prevalence of cognitive decline in older individuals with type 2 diabetes and generate data to inform future guidelines for cognitive screening and interventions in this population.

ELIGIBILITY:
Inclusion Criteria for the Prevalence Study (Cognitive Screening):

* Age ≥ 65 years
* Diagnosis of Type 2 Diabetes (T2D)
* Patient at the outpatient clinic at either Bispebjerg Hospital, Rigshospitalet, or Steno Diabetes Center Copenhagen
* Speaks and understands Danish (required for the cognitive tests)
* Informed written consent

Inclusion Criteria for the Randomized Controlled Trial (Multidomain Intervention):

* Meets all the above inclusion criteria, and at least one of the following:

  1. A diabetes-specific dementia score ≥ 7 (equivalent to a 40% increased risk of developing dementia within the next 10 years), and a SCIP or MoCA score ≥ 0.5 SD below the age- and education-adjusted norm
  2. A SCIP or MoCA score ≥ 1 SD below the age- and education-adjusted norm
  3. At least 2 out of 5 SCIP subtests with a score ≥ 1 SD below the age- and education-adjusted norm

     Exclusion Criteria for the Prevalence Study (Cognitive Screening):
* Diagnosis of dementia or prior referral to a dementia clinic
* Diagnosis of psychiatric, neurological, or other disorders that, in the investigator's opinion, hinder participation in cognitive screening, preclude compliance with the study protocol, or affect the evaluation of results

Exclusion Criteria for the Randomized Controlled Trial (Multidomain Intervention):

* Meets all the above exclusion criteria
* Participants whose cognitive MoCA screening indicates dementia will be excluded and advised to contact their physician
* Participants unwilling to engage in parts of the multidomain intervention will be excluded

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 420 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2029-06 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
Difference in Change in Cognitive Function | 2 years
  Difference in change in cognitive function (visit 1 compared to follow-up) measured by SCIP between the multifactorial intervention group and the usual care group.

SECONDARY OUTCOMES:
The Number of Hospitalizations Related to All-cause Disease | 2 years
Changes in Health-related Quality of Life Measured by SF-36 | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Jørgen Rungby, Professor, MD, DMSc, Study Chair — Steno Diabetes Center Copenhagen; Malin S.D. Nilsson, MD, PhD, Principal Investigator — Steno Diabetes Center Copenhagen
Locations (3):
- Denmark (3):
  - Department of Endocrinology, Rigshospitalet, Copenhagen
  - Department of Endocrinology, Bispebjerg-Frederiksberg Hospital, Copenhagen
  - Steno Diabetes Center Copenhagen, Herlev

IPD SHARING:
Plan to Share IPD: Undecided